CLINICAL TRIAL: NCT04087798
Title: Controlling Hypertension Through Education and Coaching in Kidney Disease
Acronym: CHECK-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Julie Wright-Nunes, Associate Professor Department of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00136011; R01DK115844-01 (NIH)
Record Dates: First submitted 2019-08-24; First posted 2019-09-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases; Chronic Disease; Chronic Kidney Disease, Stage 3 (Moderate); Chronic Kidney Disease, Stage 4 (Severe); Chronic Kidney Disease Stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Disease; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Eligible patients enrolled from the control group clinics will be given a Control-EDI which has information about kidney disease in general (not tailored to the patient) during their clinic visit.
  Interventions: Behavioral: Control-EDI
- Intervention (Experimental): Eligible patients enrolled from the intervention group clinics will be given an Intervention-EDI which has personalized information about kidney disease. There will be space on this for the provider to type in any goals or key points they want the patient to remember. Additionally, patients in this group will also receive health coaching.
  Interventions: Behavioral: Intervention-EDI and health coaching

INTERVENTIONS:
Behavioral: Control-EDI — Patients in the control group will receive Control-EDI from their primary care provider during clinic visit. Subsequent patient CKD education and follow-up will be provider dependent. Patients will be called and reminded of their study visits at 1, 6, 12 months to complete study measures, BP checks, and give urine and blood samples (baseline and 12-month visit only).
  Other Names: Control-Encounter Decision Intervention
  Arms: Control
Behavioral: Intervention-EDI and health coaching — Patients in the intervention group will receive a personalized Intervention-EDI from their primary care provider during visit, which will include their most recent BP, their urine protein level and most recent eGFR. There is also a space for their provider to type in a sentence about specific goals for the patient.
  Health coaches will conduct a baseline call and 4-6 coaching calls, based on patient's needs, over an 11-month period. There are 4 topic areas related to blood pressure and CKD that will be the focus of the calls. Coaches will also have pre-determined and vetted educational resources to provide patients if needed. Additionally, patients will be called and reminded of their study visits at 1, 6, 12 months to complete study measures, BP checks, and give urine and blood samples (baseline and 12-month visit only).
  Other Names: Intervention-Encounter Decision Intervention
  Arms: Intervention

SUMMARY:
Chronic kidney disease (CKD) is a serious and growing public health problem. The purpose of this study is to find out if an educational worksheet, called the Encounter Decision Intervention (EDI), combined with health coaching helps CKD patients improve their blood pressure and other health outcomes. The research team hypothesizes that the intervention group will have greater improvement in CKD outcomes than the control group.

DETAILED DESCRIPTION:
Patients that meet eligibility criteria and are seen in a clinic assigned to the control group will be given a Control-Encounter Decision Intervention (Control-EDI) about kidney disease in general (not tailored to the patient) by their primary care provider. Eligible patients that agree to participate and give consent will complete enrollment, 1, 6, and 12 month follow-up visits.

Eligible patients that are seen in a clinic assigned to the intervention group will be given a personalized Intervention-EDI by their primary care provider. Following this, eligible patients that agree to participate and give consent will complete the enrollment visit, and have a baseline call with a health coach. In addition to the 1, 6, 12 month follow-up visits these patients will also have approximately 4-6 phone calls with the health coach between the baseline visit and 11 months after enrollment.

In both groups the study team will be collecting medical information and assessments regarding their health; blood sample and urine samples at baseline and 12 months; approximately 4-6 phone calls; as well as surveys at various time points.

In order to reduce in-person human subject activity due to the Coronavirus disease 2019 (COVID-19) pandemic, participants in both groups receive an at home blood pressure monitor so that systolic- & diastolic-BP data can be collected at all 4 time points (baseline, 1, 6, 12 months). Additionally, we have increased the window tolerance for data collection by a few months for greater flexibility.

We also collect survey data from patients' providers to assess their perception of the intervention's usefulness after patients complete their follow-up study visits. The provider survey data collection will occur up to one year, with an anticipated 100 participating providers. In addition to the 320 patients already enrolled, the study is expected to include a total of 420 participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CKD stage 3, 4, or 5 documented in medical record
* Aware of CKD diagnosis
* Has diagnosis of hypertension documented in medical record and most recent Blood Pressure (BP) within the last year meets criteria of uncontrolled hypertension (≥140 mmHg, and/or a diastolic blood pressure ≥90 mmHg noted in an ambulatory care setting within the past one year)
* Estimated glomerular filtration rate (eGFR) of <60 within the last 18 months documented in the medical record

Exclusion Criteria:

* Currently on dialysis permanently (i.e. are considered "end-stage renal disease" and receiving dialysis)
* Previous kidney transplant
* Pregnant (indicated by medical record or if patient self-identifies as pregnant)
* Has cognitive, language, or vision impairment(s) that would prohibit participating in education, taking surveys, or participating in coaching activities
* Has terminal illness

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure between baseline and 12 months | Baseline, 12 months
  Changes in systolic blood pressure between baseline and 12 months will be compared between the intervention group and control group.

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure between baseline and 12 months | Baseline, 12 months
  Changes in diastolic blood pressure between baseline and 12 months will be compared between the intervention group and control group.
Slope of systolic BP between baseline and 12 months using all available BP values | Baseline up to 12 months
  BP will be collected at 4 time points - baseline, 1, 6, 12 months. This will be compared between the intervention group and control group.
Slope of diastolic BP between baseline and 12 months using all available BP values | Baseline up to 12 months
  BP will be collected at 4 time points - baseline, 1, 6, 12 months. This will be compared between the intervention group and control group.
CKD knowledge measured by the Kidney Knowledge Survey (KiKS) | Baseline up to 12 months
  This is a 28-item questionnaire measuring objective CKD disease knowledge and includes questions about goals, cardiovascular risk, and anti-hypertensive medications. Patients will answer the questions with a yes or no answer and their score will be based on how many responses were correct. This number will be converted to a percentage.
Medication Adherence Self-Efficacy Scale-Revised (MASES-R) | Baseline up to 12 months
  This is a 13-item measure with the answers on a Likert scale of 1 (not at all sure) to 4 (extremely sure). The higher the score the higher the self-efficacy, with a range from 13-52.
Morisky Medication Adherence Scale (MMAS - 8) | Baseline up to 12 months
  This scale is to quantify adherence to pharmacological treatments by 8 items. Levels of adherence are based on the following scores: <6 = low adherence; 6-<8 = medium adherence; 8 = high adherence.
Visit Time with provider | Enrollment visit (baseline)
  Length of time provider spends with the patient. This will be compared between the intervention group and control group.
Total time in clinic | Enrollment visit (baseline)
  Length of time between patient check-in and check-out. This will be compared between the intervention group and control group.
Patient Motivation by the Treatment Self-Regulation Questionnaire scale (TSRQ) | Baseline up to 12 months
  This contains a 17-item questionnaire in which the participants select scores from 1-7 or does not apply. A number of 1 = not at all and a score of 7 = considered very true, and zero = not applicable.
Satisfaction with CKD care based on Communication Assessment Tool (CAT) | Baseline up to 12 months
  This is a 15-item questionnaire that assesses the quality of physician to patient communication completed by the patients. There are 5 answers to choose from; poor, fair, good, very good, and excellent. The Score range is 1-5, where 1 means negative perception of communication and 5 means positive perception of communication.
Satisfaction with CKD care based on Consultation Care Measure (CCM) | Baseline up to 12 months
  This is a 21-item questionnaire that is completed by the patients, and select from the the 4 choices: very strongly agree, strongly agree, agree, and neutral/disagree.
  Each answer is worth one point on a Likert scale with a higher score meaning more satisfied.
Perceptions of health coaching for the intervention group | Baseline up to 12 months
  During health coach phone calls, participants will be asked 37 questions about their perceptions of the health coach program, including how much their participation in CHECK-D helped participants change various behaviors. Participant responses will be used to examine various measures of reliability and validity during the analyses of data acquired though this survey.
Self-efficacy for disease self-management based on The Perceived Kidney/Dialysis Self-Management Scale (PKDSMS) | Baseline up to 12 months
  This is an 8-item scale regarding self-efficacy where each statement is rated on the level of agreement from 1-5. 1 is disagree and 5 is agree.
Self-reported Blood Pressure-Related Behaviors Survey | Baseline up to 12 months
  This is a 5-item survey about knowledge and behaviors regarding sodium in the diet.
Provider Adoption based on EMR query and patient survey | Baseline
  Provider adoption will be measured by the percentage of enrolled patients whose providers used the EDI with them during their visit. Data will be collected by EMR query and a 1-item question in the patient survey.
Provider Fidelity measured by EMR query | Baseline
  Provider fidelity will be measured by the percentage of enrolled patients in the intervention clinics whose providers entered 1-2 patient specific goals in the EDI. This will be collected through EMR query.
Provider Perception of Usefulness by provider survey | After all patient follow-ups, up to one year
  Provider perception of usefulness will be measured by a survey of 2-3 questions about how useful they thought it was.
Change in serum creatinine | Baseline, 12 months
  Change in Serum Creatinine between baseline and 12-months
Change in urine protein-creatinine ratio | Baseline, 12 months
  Change in urine protein-creatinine ratio between baseline and 12-months
Change in estimated glomerular filtration rate (eGFR) | Baseline, 12 months
  Change in estimated glomerular filtration rate (eGFR) between baseline and 12-months
Change in EMR-recorded blood pressure between baseline and 12 months | Baseline up to 12 months
  Changes in blood pressure recorded in the EMR from baseline to 12 months will be compared between the intervention group and control group
Change in study visit blood pressure supplemented with EMR blood pressure if missing | Baseline up to 12 months
  Changes in blood pressure collected during study visits from baseline to 12 months will be compared between the intervention group and control group, with EMR data used to supplement missing values
Change in blood pressure using the combined dataset of all study visit and EMR blood pressure values | Baseline up to 12 months
  Changes in blood pressure from baseline to 12 months will be analyzed using a combined dataset that includes all available study visit and EMR blood pressure values

CONTACTS AND LOCATIONS:
Overall Officials: Julie Wright-Nunes, MD, Principal Investigator — University of Michigan
Locations (11):
- United States (11):
  - University of Michigan / Domino's Farms, Ann Arbor, Michigan
  - University of Michigan / Briarwood Family Medicine, Ann Arbor, Michigan
  - University of Michigan / Brighton Health Center, Brighton, Michigan
  - University of Michigan / Canton Health Center, Canton, Michigan
  - University of Michigan / Chelsea Health Center, Chelsea, Michigan
  - University Health Center - GMAP/Gen Med, Detroit, Michigan
  - University Health Center - Med Peds, Detroit, Michigan
  - University of Michigan / Dexter Health Center, Dexter, Michigan
  - University of Michigan / Livonia Health Center, Livonia, Michigan
  - University of Michigan / Northville Health Center, Northville, Michigan
  - University of Michigan / Ypsilanti Health Center, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wright Nunes JA, Resnicow K, Richardson C, Levine D, Kerr E, Saran R, Gillespie B, Bragg-Gresham J, Delacroix EL, Considine S, Fan A, Ellies T, Garcia-Guzman L, Grzyb K, Klinkman M, Rockwell P, Billi J, Martin C, Collier K, Parker-Featherstone E, Bryant N, Seitz M, Lukela J, Brinley FJ, Fagerlin A. Controlling Hypertension through Education and Coaching in Kidney Disease (CHECK-D): protocol of a cluster randomised controlled trial. BMJ Open. 2023 Aug 1;13(8):e071318. doi: 10.1136/bmjopen-2022-071318. PMID 37527897

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT04087798/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04087798/ICF_000.pdf